CLINICAL TRIAL: NCT04447508
Title: Assessing the Feasibility and Acceptability of Reframe Your Pain to Enhance Exercise Adherence in People With Chronic Low Back Pain
Brief Title: Reframe Your Pain: A Feasibility and Acceptability Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restrictions pertaining to COVD study has been halted
Sponsor: University of Manitoba (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Laura Meade, Principle Investigator,Postdoctoral Research Fellow, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2020:025
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Pain, behaviour change, exercise
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise class and motivational interviewing (Experimental): Patients receiving the intervention will be enrolled in an online instructor led group exercise class and five online one on one motivational interviewing sessions.
  Interventions: Behavioral: Participants receive one on one motivational interviewing and participate in a group exercise class virtually.
- Usual care (No Intervention): Participants in the control group will receive an exercise booklet and educated on the benefits of exercise for low back pain. They will be advised to exercise for the duration of the study

INTERVENTIONS:
Behavioral: Participants receive one on one motivational interviewing and participate in a group exercise class virtually. — Participants have one group exercise class over zoom per week and an online one on one motivational interviewing session every second week.
  Arms: Exercise class and motivational interviewing

SUMMARY:
The study will follow guidelines provided by the ORBIT model for developing behavioural treatments. This model proposes that to optimize an intervention's effectiveness, its development should be undertaken in four phases. Phase 1 (design) and 2a (proof of concept) were completed during the applicant's PhD. The study will complete phase 2b (pilot-feasibility study) of the model with the aim to determine pre-defined feasibility outcomes to inform future progression to phase 3 (efficacy trial) and 4 (effectiveness trials).

DETAILED DESCRIPTION:
Approximately one in five Canadians suffer from persistent low back pain (PLBP). Experiencing PLBP limits an individual's independence by impacting their ability to participate in family, social and working life. Canada has the second highest rate of opioid prescribing in the world and this comes with many risks, including an increase in admissions to addiction programs and opioid related deaths. Due to the widespread economic, personal and social impacts, World Health Organization burden of disease profiles have shifted focus from the treatment of communicable disease to the treatment of non-communicable, long term diseases, including non-pharmaceutical treatment of PLBP.

Active treatment, including physical activity and exercise has been shown to effectively reduce pain severity while increasing function and quality of life in patients with PLBP. However, over half of the patients that are prescribed exercises as treatment for their conditions do not adhere and there is a recognized gap in the literature of research exploring exercise adherence in this population.

Preliminary work in this research program included the development and initial testing of a behaviour change intervention to enhance exercise adherence in a population PLBP. Using the intervention development framework Intervention Mapping, a group-based exercise program incorporating an exercise app and one on one psychological support was developed. However, assessment within a Canadian context, its clinical significance and efficacy for wider implementation have not yet been assessed.

The primary objective of the proposed project is to inform progression to a large scale randomized controlled trial of the intervention (vs usual care) through the evaluation of a pilot-feasibility trial and an efficacy trial.The study will employ a two-arm randomized controlled pilot-feasibility study with a nested qualitative interview study.

The purpose of pilot-feasibility trials is to assess feasibility of a protocol to provide estimates for an efficacy trail. Therefore, while the design may look similar to an efficacy trial, clinical outcomes are not the primary outcome. Due to their smaller sample size, pilot-feasibility studies may provide unstable estimate of effect size, however their assessment will determine the sample size needed for the efficacy trial. This study will allow for the feasibility of transferring the program from a UK context (where it was originally tested) to a Winnipeg setting.

The program offered will be delivered to patients with PLBP as an adjunct to physiotherapy designed to facilitate self-management to enhance exercise adherence. Patients receiving the intervention will be asked to complete an online instructor led group exercise class and five online one on one motivational interviewing sessions.

Objectives:

The primary objectives of the study are to:

(i) determine feasibility of recruitment (ii) determine adherence to study protocol (iii) determine completion rates of outcome measures (iv) provide parameters needed for sample size calculations for future research

Methods Participants will be recruited through the Spine Assessment Clinic at the Health Sciences Centre and the study will be conducted at the Reh Fit Centre. The signed informed consent form will be collected at the baseline meeting and baseline measures collected. Participants will then be randomised to the intervention or control group (computer generated). Allocation will be single blinded as the personnel delivering the intervention will be aware of who is in the intervention group. However an independent researcher (research assistant) will collect and anonymise the data prior to analyses.

All participants will be provided with the exercise program booklet and exercise diary. Control participants will be asked to compete the exercises twice a week. Intervention participants will be scheduled for their motivational interviewing sessions and enrolled in the exercise program.

Participants randomised to the intervention will be enrolled in the group exercise class. The class will be a rolling start, so that participants will start the exercise class once enrolled in the study and finishing after six weeks. Therefore, not all participants will start at the same time to avoid some participants waiting for a long duration until 10 participants are randomised to the intervention group. The exercise class will be one hour in duration and run once a week for 6 weeks. It will be conducted virtually using Zoom.

Four motivational interviewing sessions will be provided concurrently with the group exercise class and held over Zoom. Motivational interviewing is a person-centered form of communication to support behaviour change. These sessions, informed by behaviour change theory, employ motivational techniques guided by the motivational interviewing protocol. The sessions are typically 30-45 minutes in duration and guided by the needs of the participant, however to inform progress and training, a guideline has been previously created during the applicant's PhD to ensure behaviour change methods are being utilised. The first session will occur at the start of the intervention with the duration between each appointment doubling each time. Following completion of the exercise class participants will be asked to attend a final online (Zoom) follow up motivational interviewing sessions at six weeks post intervention. The content of this session will be similar to the previous sessions and driven by the participant, however will be to assess the self-management techniques the participant may or may not have used to continue to engage with their exercises on their own. Zoom is an encrypted software that allows for secure web conferencing. Health support provided by e-health programming is becoming more prominent in the literature and promotes accessibility and cost-effectiveness to care. Motivational interviewing has been provided to patients with persistent pain and its delivery within this context is warranted.

Following completion of the final follow up, participants will be invited to complete a qualitative interview with researchers to assess acceptability of the intervention, as well as to explore personnel most appropriate to deliver motivational interviewing. Staff involved in delivering the intervention will also be invited to provide their views of acceptability of intervention implementation. The interview topic guides will be informed by the Theoretical Framework of Acceptability which outlines seven constructs to assess program acceptability; ethicality, affective attitude, burden, opportunity costs, perceived effectiveness, self-efficacy, and intervention coherence. These interviews will be conducted by an independent researcher (research assistant) to facilitate open and honest responses by the participants.

Following the acceptability interviews participants will be debriefed on the study. This will take approximately 5 minutes and the research assistant will share with the participant the rationale and purpose of the study and explain which group they were randomised to. For control participants this will take place following their completion of the final questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years old)
* Low back pain for three months or longer and no current plans for surgical intervention
* Previously been prescribed exercises by a physiotherapist

Exclusion criteria:

* Plans for long absences during the study period
* Participating in other studies or interventions targeting exercise or behaviour change during study
* Recent (2 months) changes to medications
* Receiving or have received prior psychological interventions for their pain (i.e., cognitive behavioural therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Eligibility | Through study completion, up to 12 weeks
  Number of eligible participants identified/week
Recruitment | Through study completion, up to 12 weeks
  Percentage of eligible participants recruited/week
Treatment completion | Through study completion, up to 12 weeks
  Percentage of participants that complete at least 3 of 5 motivational interviewing sessions and 5 of the 6 exercise classes
Follow up | Through study completion, up to 12 weeks
  Loss of follow up at 6 weeks post intervention
Completion of outcome measures | Through study completion, up to 12 weeks
  Percentage of participants that complete baseline and follow up measures and complete exercise diary

SECONDARY OUTCOMES:
Exercise adherence rating scale (EARS) | Baseline, 6 weeks, 12 weeks
  16 item questionnaire on 5-point Likert scale (0-completely agree, 4-completely disagree) higher scores indicating stronger adherence to exercise.
Optimal Screening for Prediction of Referral and Outcome (OSPRO) questionnaire | Baseline, 6 weeks, 12 weeks
  17 item questionnaire to determine yellow flags to outcomes. Domains measured include negative mood, fear-avoidance, positive affect/coping. Higher scores equate to better outcomes.
Musculoskeletal health (MSK-HQ) | Baseline, 6 weeks, 12 weeks
  14 item questionnaire to measure constructs of pain and function. The item is scored on a range of 0-56, with a better score indicating better MSK-HQ health status. The total score is calculated by adding the numbers next to the box that the respondent has ticked on the questionnaire form.
Health Action Process Approach (HAPA)constructs | Baseline, 6 weeks, 12 weeks
  Measures domains of outcome expectations,risk perception,self-efficacy, action and coping plans; the variables of the theoretical model underpinning the intervention. Each domain has one question with 5 anchor points on a 4 point Likert scale (0-not true at all, 4-Exactly true). Higher scores indicate stronger strong use of the concepts. A change in scores will indicate if the intervention targeted the concepts it is theorized to target.
Exercise adherence self report | Through study completion, up to 12 weeks
  Exercise log

IPD SHARING:
Plan to Share IPD: Undecided
Feasibility outcomes may be shared with other researchers to inform progression in other parallel research

REFERENCES:
- [Background] Summers S. Evidence-based practice part 1: pain definitions, pathophysiologic mechanisms, and theories. J Perianesth Nurs. 2000 Oct;15(5):357-65. doi: 10.1053/jpan.2000.18211. PMID 11811340
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Briggs AM, Woolf AD, Dreinhofer K, Homb N, Hoy DG, Kopansky-Giles D, Akesson K, March L. Reducing the global burden of musculoskeletal conditions. Bull World Health Organ. 2018 May 1;96(5):366-368. doi: 10.2471/BLT.17.204891. Epub 2018 Apr 12. No abstract available. PMID 29875522
- [Background] Gomes T, Mamdani MM, Dhalla IA, Cornish S, Paterson JM, Juurlink DN. The burden of premature opioid-related mortality. Addiction. 2014 Sep;109(9):1482-8. doi: 10.1111/add.12598. Epub 2014 Jul 7. PMID 25041316
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Meade LB, Bearne LM, Sweeney LH, Alageel SH, Godfrey EL. Behaviour change techniques associated with adherence to prescribed exercise in patients with persistent musculoskeletal pain: Systematic review. Br J Health Psychol. 2019 Feb;24(1):10-30. doi: 10.1111/bjhp.12324. Epub 2018 Jun 17. PMID 29911311
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Kok G, Gottlieb NH, Peters GJ, Mullen PD, Parcel GS, Ruiter RA, Fernandez ME, Markham C, Bartholomew LK. A taxonomy of behaviour change methods: an Intervention Mapping approach. Health Psychol Rev. 2016 Sep;10(3):297-312. doi: 10.1080/17437199.2015.1077155. Epub 2015 Oct 15. PMID 26262912
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083